CLINICAL TRIAL: NCT06164405
Title: RESPONSE OF ARTERIAL dP/dt TO FLUIDS AND VASOACTIVE DRUGS DURING ABDOMINAL SURGERY: A PROSPECTIVE PILOT STUDY
Brief Title: Arterial dP/dt Dependency on Loading Conditions
Acronym: REABILITY
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RUSSO ANDREA, medical doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6166
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Intraoperative Hemodyamic Monitoring
Keywords: emodinamica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: arterial dp/dtmax — to assess the variations of the arterial dp/dt max after drugs or fluids administration

SUMMARY:
In the present study the investigators aim to assess the changes of the arterial dP/dtmax induced by fluids and vasoactive drugs during abdominal surgery

ELIGIBILITY:
Inclusion Criteria:

patients scheduled for abdominal surgery informed consent acceptance

-

Exclusion Criteria:

* BMI> 30 Kg /m2;
* Atrial Fibrillation;
* Congestive heart failure with FE <35% and/or NYHA≥3;
* Severe known cardiac valve disease;
* Emergency surgery
* Shock or any acute conditions who required admission intensive care unit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: surgical patients
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
dp/dt fluids dependency | intraoperative
  measurement of dp/dtmax after fluid challenge

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitairo Agostino Gemelli, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No